CLINICAL TRIAL: NCT01141036
Title: Propofol Versus Midazolam for Upper Endoscopy in Cirrhotic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Liver Clinic, Ziv medical center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 006-08; 006-08ziv
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Cirrhosis
Keywords: Propofol; Midazolam; sedation; cirrhosis; endoscopy; recovery time; efficacy and safety of sedation; patient satisfaction; return to baseline function; saturation of oxygen
MeSH Terms: conditions — Fibrosis; Patient Satisfaction | interventions — Propofol; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol (Active Comparator): propofol
  Interventions: Drug: propofol
- Midazolam (Active Comparator): Midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: propofol — Propofol will be initiated with a 30-50 mg i.v. bolus followed by repeated 10-20 mg doses at variable intervals (approximately 15 s, at the discretion of the endoscopist/nurse) until an appropriate level of sedation will be achieved.
  Arms: propofol
Drug: Midazolam — Midazolam (0.5-1.0 mg) will be administered in a similar fashion with incremental dosing at intervals of approximately 1-3 min until a level of sedation will be achieved
  Arms: Midazolam

SUMMARY:
Upper GI endoscopy is often performed in patients with chronic liver disease to screen for esophageal and gastric varices. The purpose of this study is to compare propofol to midazolam for sedation in patients with chronic liver disease undergoing diagnostic upper GI endoscopy.

DETAILED DESCRIPTION:
Background : Upper GI endoscopy is often performed in patients with chronic liver disease to screen for esophageal and gastric varices. AIM: The purpose of this study is to compare propofol to midazolam for sedation in patients with chronic liver disease undergoing diagnostic upper GI endoscopy. Methods: 60 outpatients who has known chronic liver disease (Child-Pugh class A or B) (cirrhosis) and are undergoing variceal screening will be randomized to receive propofol or midazolam for sedation. Administration of sedation was performed by a anesthesist. Outcome measures studied are induction and recovery times, efficacy and safety of sedation, patient satisfaction, and return to baseline function and subclinical hepatic encephalopathy (number connection test), and saturation of oxygen. expected results: The mean time to achieve adequate sedation will be shorter for for the propofol group in comparison to midazolam group. The level of sedation achieved by the propofol group will be greater. Time to full recovery will be faster in the propofol group. Propofol do not exacerbate subclinical hepatic encephalopathy as compared to midazolam. patients receiving propofol will express greater overall mean satisfaction with the quality of their sedation at the time of discharge. Conclusions: Propofol sedation is expected not to exacerbate subclinical hepatic encephalopathy in cirrhotics.

ELIGIBILITY:
Inclusion Criteria:

* Known chronic liver disease (Child-Pugh class A or B) who presented for upper GI endoscopy for routine variceal screening.
* The diagnosis of liver disease will be based on available past history, serological testing, radiological imaging, and liver histology when available.
* Staging of cirrhosis will be determined by MELD score and by Child-Pugh score . All patients will complete a standard preprocedure history and physical examination to establish current degree of encephalopathy and ascites.

Exclusion Criteria:

* Exclusion criteria will include the following:

  * known allergy or adverse reaction to sedative or component thereof
  * patients with known significant respiratory disease or airway abnormality)
  * active neurological impairment including clinically detectable hepatic encephalopathy
  * advanced or decompensated liver disease ( CP score >10, MELD >24) (Child-Pugh class C)
  * active alcohol consumption or illicit drug abuse
  * active prescription for sedation or narcotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Exacerbation of hepatic encephalopathy

SECONDARY OUTCOMES:
Recovery time, time to discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv medical center liver unit, Safed, Israel, Israel